CLINICAL TRIAL: NCT00221572
Title: Can Quantitative Ultrasound be Used for the Evaluation of Bone Health in Adolescents and Adults With Cystic Fibrosis
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: 2005/149
Record Dates: First submitted 2005-09-12; First posted 2005-09-22 (Estimated); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Determination of bot density of Cystic Fibrosis patients — Determination of bot density of Cystic Fibrosis patients.

SUMMARY:
Measurement of bone density of Cystic Fibrosis patients with two techniques and correlation to serum bone parameters, use of steroids, lung function and nutritional status.

DETAILED DESCRIPTION:
Measurement of bone density of Cystic Fibrosis patients with two techniques and correlation to serum bone parameters, use of steroids, lung function and nutritional status.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Cystic Fibrosis

Exclusion Criteria:

-

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Cystic Fibrosis
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2006-06 (Actual); Primary Completion 2011-06-16 (Actual); Study Completion 2011-06-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Van Biervliet, MD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website University Hospital Ghent — http://www.uzgent.be